CLINICAL TRIAL: NCT04771507
Title: A Pilot Study on Intermittent and Repeated Dosing of Ibrutinib in the Treatment of Patients With Advanced-phase Chronic Lymphocytic Leukemia (CLL)
Brief Title: A Pilot Study on Intermittent Ibrutinib in Patients With Advanced-phase Chronic Lymphocytic Leukemia (CLL)
Acronym: IbruOnOff
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jeanette Lundin (Other)
Responsible Party: Sponsor-Investigator, Jeanette Lundin, Consultant, Associate Professor, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCK-LT-CLL02/2017
Record Dates: First submitted 2021-02-19; First posted 2021-02-25 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ibrutinib

STUDY DESIGN:
Intervention Model Description: Patients treated with ibrutinib for at least 6 months and have achieved at least partial response will after inclusion stop the ibrutinib treatment and be followed-up for the study. If progress, they will re-initiate ibrutinib treatment. When they achieve at least partial response they stop the treatment again, and so on.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intermittent ibrutinib (Experimental): Intermittent treatment with ibrutinib.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib will be stopped at inclusion in the and the patient will be followed OFF therapy. At clinical progress, ibrutinib will be restarted (ON period) at the same standard dose as used at inclusion. When the patient achieve at least partial response again, a new OFF period is started, and so on.
  Other Names: Imbruvica

SUMMARY:
Ibrutinib, an inhibitor of Bruton´s tyrosine kinase (BTK) is approved in CLL as continuous, daily administration of 420 mg orally until progression. Ibrutinib drug costs in health care are rapidly increasing and are difficult to predict, as long-term follow up analyses have shown that many patients remain on therapy for several years, in some cases even many years. It has been observed that patients who stop ibrutinib due to side effects may often remain with continued CLL disease control i.e. in stable partial remission even when off ibrutinib therapy. There are also emerging data on mutations within BTK, with loss of efficacy of ibrutinib, during long-term continuous administration. These observations raise the question whether alternative dosing strategies may be feasible. This pilot study will explore intermittent and repeated dosing of ibrutinib, until alternative therapy is required due to resistance or intolerance to ibrutinib. An "ON-OFF" dosing strategy will be applied, where advanced-phase CLL patients who have received at least 6 months of ibrutinib and who have achieved a stable PR will stop ibrutinib and be followed off therapy until clinical progression, at which ibrutinib will be re-instituted. Such "ON-OFF" ibrutinib cycles may be repeated until non-tolerability or resistance, or need of continuous dosing of ibrutinib (i.e. early progression when off the drug). If successful, the study will indicate a way forward towards reducing ibrutinib drug costs in health care without affecting long-term disease control, possibly also with fewer ibrutinib-related side effects due to a lower cumulative dose of ibrutinib. Long-term effects on potential mutations within BTK and its downstream signaling molecules will also be analysed.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and voluntarily provide written informed consent and comply with the requirements of the study.
2. Age 18 years and older. There is no upper age limit in this trial.
3. Able to adhere to the study visit schedule and other protocol requirements.
4. Before start ibrutinib for the first time: diagnosed with CLL/SLL and active disease in need of treatment after having failed chemoimmunotherapy for CLL defined as a) refractory according to iwCLL criteria; or b) relapsed and deemed not suitable for additional chemo- or chemoimmunotherapy or c) del 17p and/or TP53 mutation irrespective of prior therapy.
5. Having received at least 6 months of ibrutinib therapy and having achieved at least clinical PR according to IWCLL criteria.
6. ECOG performance status of </= 2 at screening.
7. Laboratory test results:

   * Absolute neutrophil count >/= 0.5 x 109/L
   * Platelet count >/= 30 x 109/L
   * Serum creatinine < 177 µmol/L
   * ASAT (SGOT) and ALAT (SGPT) >/= 2 x ULN or >/= 5 x ULN unless attributable to CLL/SLL
8. Disease free of prior malignancies for >/= 2 years with exception of currently treated basal cell, squamous cell carcinoma of the skin, or carcinoma "in situ" of the cervix or breast.
9. Agree to use reliable forms of contraception. Post-menopausal females and surgically sterilized females are exempt from this criterion.

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or breast feeding females.
3. Any condition, including the presence of laboratory abnormalities, which according to the responsible physician places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study.
4. Use of any other experimental therapy within the last 14 days.
5. Concurrent use of other anti-cancer agents or treatments than ibrutinib (except a low dose of corticosteroids, max 10 mg of prednisone/day).
6. Positivity for HIV or infectious hepatitis, type A, B or C.
7. Opportunistic infections within the last 3 months.
8. Patient planned for or being a potential candidate for allo-SCT.
9. Uncontrolled hemolytic anemia or autoimmune thrombocytopenia.
10. CNS involvement or history of Richter's transformation.
11. Requires or has received anticoagulation treatment with warfarin or equivalent Vitamin K antagonists (eg, phenprocoumon) within 28 days of the first dose of ibrutinib.
12. Requires treatment with a strong cytochrome P450 (CYP) 3A4/5 inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-02-23 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety measured as type, frequency and severity of adverse events. | Through study completion, 1-24 months.
  Type, frequency and severity of adverse events and relationship to intermittent ibrutinib dosing.

SECONDARY OUTCOMES:
Overall response at each treatment cycle. | Through study completion, 1-24 months.
  Response when re-starting ibrutinib, at each cycle.
Time to PR and PR-L at each cycle. | Through study completion, 1-24 months.
  Time to partial response (PR) and partial response with persistent lymphocytosis (PR-L) when re-starting ibrutinib, at each cycle.
Time to stop until restart of ibrutinib due to progress | Through study completion, 1-24 months.
  Time from the patient going off ibrutinib until it has to be re-started due to progressive, for each cycle.disease (PD), at each cycle.
Number of ibrutinib treatment cycles and OFF therapy periods. | Through study completion, 1-24 months.
  The number of cycles each patient stop and re-start ibrutinib.
Cumulative dose of ibrutinib. | Through study completion, 1-24 months.
  The cumulative dose of ibrutinib for each patient.
Overall survival. | Through study completion, 1-24 months.
  Overall survival.
Risk of early rebound phenomenon. | Through study completion, 1-24 months.
  Observation of early rebound phenomemon at each re-start of ibrutinib.
Time to need of alternative treatment. | Through study completion, 1-24 months.
  Time to need of alternative treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette Lundin, MD PhD, Principal Investigator — Karolinska University Hospital
Locations (9):
- St Olavs Hospital, Trondheim, Norway
- Sweden (8):
  - Falu lasarett, Falun, Dalarna County
  - Gävle Hospital, Gävle, Gävleborg County
  - Skåne University Hospital, Lund, Skåne County
  - Sahlgrenska University Hospital, Gothenburg
  - Örebro University Hospital, Örebro
  - Karolinska University Hospital, Stockholm
  - Norrland's University Hospital, Umeå
  - Akademiska hospital, Uppsala